CLINICAL TRIAL: NCT00352768
Title: SME3110 (Fluvoxamine Maleate) in the Treatment of Obsessive-Compulsive Disorder: A Post-marketing Clinical Study in Children and Adolescents (8 Through 18 Years of Age) -A Double-blind, Randomized, Placebo-controlled Study
Brief Title: Fluvoxamine Maleate in the Treatment of Obsessive-Compulsive Disorder: A Post-marketing Clinical Study in Children and Adolescents
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was prematurely terminated (26 June 2009) due to slow recruitment
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S114.3.118
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Fluvoxamine Maleate; OCD; Children and Adolescents
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- F (Experimental)
  Interventions: Drug: Fluvoxamine maleate
- P (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine maleate — Test product: Fluvoxamine maleate 25mg tablet. In case that the daily dose is one tablet, the study medication will orally be administered once daily, at bedtime. In case that the daily dose is two tablets or higher (maximam:6 tablets), the study mmedica
  Arms: F
Drug: Placebo — Placebo
  Arms: P

SUMMARY:
This study is to verify the efficacy of fluvoxamine maleate given for 10 weeks in treatment of children and adolescents with obsessive-compulsive disorder

ELIGIBILITY:
Inclusion Criteria Have a minimum total score of 16 on the JCY-BOCS, Weight is within the standard weight ± 2S.D. based on the standard weight for each age in the School Health Statistical Survey Exclusion Criteria Have the following predominant psychiatric diagnosis -Schizophrenia Have previously been treated with fluvoxamine maleate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
the time of onset of 25% decrease from baseline in the Japanese Version of the Children's Yale-Brown Obsessive Compulsive Scale (JCY-BOCS) 10-item total score | 10 weeks

SECONDARY OUTCOMES:
The Clinical Global Impression(CGI) improvement at Week 10 | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshiaki Yamaguchi, Study Director — Solvay Pharmaceuticals
Locations (11):
- Japan (11):
  - S114.3.118 Kohnodai Hospital, National Center of N, Chiba Prefecture
  - S114.3.118 Kyushu University Hospital, Fukuoka Prefecture
  - S114.3.118 Hiroshima-city Funairi Hospital, Hiroshima Prefecture
  - S114.3.118 Goryokai Hospital, Hokkaido Prefecture
  - S114.3.118 Hyogo Children's Hospital, Hyogo Prefecture
  - S114.3.118 Kobe University Hospital, Hyogo Prefecture
  - S114.3.118 National Hospital Organization Kagawa C, Kagawa Prefecture
  - S114.3.118 National Hospital Organization Kikuti N, Kumamoto Prefecture
  - S114.3.118 National Hospital Organization Sakakiba, Mie Prefecuture
  - S114.3.118 Nara Medical University Hospital, Nara Prefecture
  - S114.3.118 Tokushima University Hospital, Tokushima Prefecture